CLINICAL TRIAL: NCT06434181
Title: Beetroot Juice for Boosting Immunity During a Time of Stress.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Baylor University (Other)
Collaborators: Southern Methodist University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 1866308
Record Dates: First submitted 2024-05-20; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The lead researcher, data collectors, and participants were blinded to the conditions. The distribution of the supplements for each condition was performed by a member of the staff that was not involved with the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beetroot Juice (Experimental): Participants in this group are given 7 daily doses of a dietary nitrate supplement (Beet-it Sport beetroot juice shots, ) and asked to drink two doses daily during the week of their final academic examinations of that term in college.
  Interventions: Dietary Supplement: Beetroot Juice
- Placebo Control (Placebo Comparator): Participants in this group are given 7 daily doses of a placebo matched in appearance and taste (Beet-it Sport placebo juice shots) and asked to drink two doses daily during the week of their final academic examinations of that term in college.
  Interventions: Dietary Supplement: Placebo Control

INTERVENTIONS:
Dietary Supplement: Beetroot Juice — Beet-It Sports Shot, 70mL, containing 6.5 mmol nitric oxide (taking two shots per day in active group)
  Arms: Beetroot Juice
Dietary Supplement: Placebo Control — Beet-It Placebo Shot, 70mL (taking two shots per day in placebo group)
  Arms: Placebo Control

SUMMARY:
The purpose of the present study is to explore the effects of a dietary nitrate supplement (i.e., beetroot juice) on nitric oxide levels, immunity, mood, and cardiovascular activity during and following final exam stress in healthy individuals.

DETAILED DESCRIPTION:
Research has demonstrated that during times of high stress (i.e., during final exam period), there is a decrease in fraction of exhaled nitric oxide (FeNO) in healthy undergraduate students. Additionally, a separate line of research has demonstrated periods of high stress impact immunity and the cardiovascular system. Nitric oxide may have a benefit in improving the physiological and psychological consequences of stress.

The present research aims to explore the impact of a dietary supplement (beetroot juice drink) on immunity, nitric oxide levels, cardiovascular activity, and mood during and following final exam stress. In this study, investigators monitor changes in cold symptoms, IL-8, blood pressure, airway nitric oxide, and mood in students during the time of final exams and a comparable time of low stress during the term. There are three laboratory assessment visits, as well as a brief questionnaire on a separate day. During the final exam period, half of the participants are randomly assigned to the experimental group provided with a dietary supplement (beetroot juice drink) of which they are asked to take two doses every day (one in the morning and one in the evening) for seven days. The other half of the participants are randomly assigned to the placebo control group provided with a placebo supplement (placebo drink) of which they are asked to take two doses every day (one in the morning and one in the evening for seven days). For the final exam period, the first of the two sessions takes place early in the examination period (first half), and the second assessment takes place in the later exam period (second half). The online questionnaire assessing symptoms is measured 3 days after the final examination period.

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled at Baylor University or Southern Methodist University

Exclusion Criteria:

* Current smoker
* Clinically significant asthma, COPD, Emphysema, heart disease, cerebrovascular disease, thyroid dysfunction, out of control diabetes
* Pregnancy, diagnosis of schizophrenia, psychosis, mood disorder, psychosis, drug or alcohol dependance

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 114 (Actual)
Dates: Start 2022-04-11 (Actual); Primary Completion 2022-12-13 (Actual); Study Completion 2022-12-13 (Actual)

PRIMARY OUTCOMES:
Wisconsin Upper Respiratory Symptom Survey (WURSS) | Baseline (non-stress mid point of semester), 1-3 days into active beetroot shots (during final examination period), 4-6 days into active beetroot shots (during final examination period), 1-3 days after finishing beetroot shots (after final examinations)
  Assesses symptoms of acute upper respiratory tract infections (common cold symptoms) by questionnaire
Changes in IL-8 levels | Baseline (non-stress mid point of semester), 1-3 days into active beetroot shots (during final examination period), 4-6 days into active beetroot shots (during final examination period)
  Change in IL-8 levels

SECONDARY OUTCOMES:
Resting blood pressure | Baseline (non-stress mid point of semester), 1-3 days into active beetroot shots (during final examination period), 4-6 days into active beetroot shots (during final examination period)
  Resting blood pressure (systolic and diastolic)
Acute stress | Baseline (non-stress mid point of semester), 1-3 days into active beetroot shots (during final examination period), 4-6 days into active beetroot shots (during final examination period)
  Perceived Stress Scale
Change in negative affect | Baseline (non-stress mid point of semester), 1-3 days into active beetroot shots (during final examination period), 4-6 days into active beetroot shots (during final examination period)
  PANAS negative affect scale
Adherence monitoring (feasibility ) | Every day, twice a day during active beetroot
  Participants will upload a cell phone video of their intake for that day to a secure cloud folder, time stamp in comparison to assigned intake windows provides measure of adherence
Exhaled Nitric Oxide | Baseline (non-stress mid point of semester), 1-3 days into active beetroot shots (during final examination period), 4-6 days into active beetroot shots (during final examination period)
  The Fraction of NO in Exhaled Breath (FENO, in ppb) will be measured with an electrochemical gas analyzer (NIOX vero).
Change in depressive symptomology | Baseline (non-stress mid point of semester), 1-3 days into active beetroot shots (during final examination period), 4-6 days into active beetroot shots (during final examination period)
  Hospital Anxiety and Depression Scale

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Southern Methodist University, Dallas, Texas
  - Annie T. Ginty, Waco, Texas

IPD SHARING:
Plan to Share IPD: Undecided